CLINICAL TRIAL: NCT00688259
Title: Cognitive-Behavioral Therapy in Veterans With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHBB-016-07S
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Results first posted 2017-12-14 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: clinical trials; psychotherapy
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Palliative Care; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Behavioral Therapy for Psychosis (CBTp) (Experimental): approximately 6 months of weekly individual manualized cognitive-behavioral psychotherapy for psychosis in which participants set personal goals, identify problematic/ illness-related beliefs and experiences that may interfere with achieving those goals, evaluate the data supporting those beliefs, and then modify the beliefs or behavior as warranted by the data to make progress on those goals.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Psychosis (CBTp)
- Supportive Therapy (ST) (Active Comparator): approximately 6 months of weekly manualized supportive psychotherapy to promote a strong alliance between the therapist and the participant in order to provide a safe place to discuss issues pertaining to the participants' lives and concerns
  Interventions: Behavioral: Supportive Therapy (ST)

INTERVENTIONS:
Behavioral: Supportive Therapy (ST) — approximately 20 sessions of manualized psychotherapy to promote a strong alliance between the therapist and the participant in order to provide a safe place to discuss issues pertaining to recovery
  Arms: Supportive Therapy (ST)
Behavioral: Cognitive Behavioral Therapy for Psychosis (CBTp) — approximately 20 sessions of individual manualized psychotherapy in which participants are taught to evaluate the data supporting beliefs that may interfere with recovery
  Arms: Cognitive Behavioral Therapy for Psychosis (CBTp)

SUMMARY:
This is a study comparing the benefits of two types of individual psychotherapy (cognitive-behavioral therapy for psychosis and supportive therapy) in symptomatic Veteran outpatients diagnosed with schizophrenia or schizoaffective disorder. Treatment lasted approximately 6 months, with outcome data on symptoms, functioning, and distress levels collected at baseline, post-treatment, and 6 months post -treatment follow-up.

DETAILED DESCRIPTION:
This is a randomized controlled trial comparing 6 months of participation in one of two active treatments, cognitive-behavioral therapy for psychosis or supportive therapy in symptomatic Veterans diagnosed with schizophrenia or schizoaffective disorder who are still symptomatic. Assessments of clinical status and social functioning were obtained at baseline, end of treatment, and 6 month follow-up. We hypothesized that participation in the cognitive-behavioral therapy would lead to greater reductions in symptoms and distress about symptoms, and more improvements in social functioning.

ELIGIBILITY:
Inclusion Criteria:

* outpatients with schizophrenia or schizoaffective disorder in proximity to the West Los Angeles VAMC
* at least one month since last hospitalization
* stable antipsychotic medication with persisting psychotic symptoms with at least minimal distress
* competent to sign informed consent.

Exclusion Criteria:

* in other individual psychotherapy
* presence of organic brain disease
* mental retardation
* illness that would prohibit regular attendance in therapy
* substance dependence diagnosis in the past 6 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2009-04; Primary Completion 2014-09 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shirley M. Glynn, PhD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data on major outcomes can be shared. Investigators can contact PI.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 122 individuals consented for study; 34 did not meet study criteria after more careful screening during baseline phase or withdrew before baseline assessments were completed; Remaining 88 were randomized.
Groups:
- Cognitive-behavioral Therapy for Psychosis (CBTp): approximately 6 months of weekly individual manualized cognitive-behavior for psychosis psychotherapy in which participants are taught to set personal goals, identify problematic beliefs and experiences that may interfere with achieving those goals, evaluate the data supporting those beliefs, and then modify the beliefs or behavior as warranted by the data to make progress on those goals.
  CBTp: approximately 20 sessions of individual manualized psychotherapy in which participants are taught to evaluate the data supporting beliefs that may interfere with recovery
- Supportive Therapy (ST): approximately 6 months of weekly manualized supportive psychotherapy to promote a strong alliance between the therapist and the participant in order to provide a safe place to discuss issues pertaining to the participants' life and concerns
  ST: approximately 20 sessions of manualized psychotherapy to promote a strong alliance between the therapist and the participant in order to provide a safe place to discuss issues pertaining to recovery
Period: Overall Study
Arm/Group | Cognitive-behavioral Therapy for Psychosis (CBTp) | Supportive Therapy (ST)
Started | 44 | 44
End to Active Treatment, (Approximately 6 months post-randomization) | 35 | 37
Completed (6 month post treatment follow-up) | 37 | 36
Not Completed | 7 | 8
Not completed — Lost to Follow-up | 2 | 4
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Declined Interview | 2 | 3
Not completed — Hospitalized at Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cognitive Behavioral Therapy for Psychosis (CBTp): approximately 6 months of weekly individual manualized cognitive-behavior for psychosis psychotherapy in which participants are taught to set personal goals, identify problematic beliefs and experiences that may interfere with achieving those goals, evaluate the data supporting those beliefs, and then modify the beliefs or behavior as warranted by the data to make progress on those goals.
  CBTp: approximately 20 sessions of individual manualized psychotherapy in which participants are taught to evaluate the data supporting beliefs that may interfere with recovery
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Therapy for Psychosis (CBTp) | Supportive Therapy (ST) | Total
Number analyzed (Participants) | 44 | 44 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.25 (9.31) | 49.07 (9.63) | 49.66 (9.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 42 | 40 | 82
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African- American | 25 | 24 | 49
  Caucasian | 11 | 15 | 26
  Asian/Pacific Islander | 3 | 2 | 5
  Latino/Hispanic | 5 | 3 | 8
Number of years since first began experiencing symptoms (self-report) [Mean (Standard Deviation); unit: years] | 24.89 (10.30) | 23.22 (11.65) | 24.06 (10.99)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Positive Schizophrenia Symptoms
Description: Mean positive symptoms Interview rating on the Brief Psychiatric Rating Scale (Ventura, Lukoff. Nuechterlein. Liberman, Green, & Shaner, 1993), with range of 1-7 and higher scores indicating greater symptoms
  Ventura, J. Lukoff D, Nuechterlein KH, Liberman RP, Green M, Shaner A: Appendix 1: Brief Psychiatric Rating Scale (BPRS) Expanded Version (4.0) scales, anchor points and administration manual. International Journal of Methods in Psychiatric Research 1993; 3:227-243
Time Frame: Pre-treatment to end of treatment, approximately 6 months post-randomization
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Cognitive-behavioral Therapy for Psychosis (CBTp): approximately 6 months of weekly individual manualized cognitive-behavioral psychotherapy for psychosis in which participants set personal goals, identify problematic/ illness-related beliefs and experiences that may interfere with achieving those goals, evaluate the data supporting those beliefs, and then modify the beliefs or behavior as warranted by the data to make progress on those goals.
  CBTp: approximately 20 sessions of individual manualized psychotherapy in which participants are taught to evaluate the data supporting beliefs that may interfere with recovery
Arm/Group | Cognitive-behavioral Therapy for Psychosis (CBTp) | Supportive Therapy (ST)
Number analyzed (Participants) | 37 | 37
units on a scale
  Baseline | 3.21 (.14) | 3.30 (.14)
  End-of-Active Treatment | 3.04 (.15) | 2.89 (.15)
Statistical Analysis 1: Comparison: Cognitive-behavioral Therapy for Psychosis (CBTp) vs Supportive Therapy (ST); Test type: Superiority or Other; p = .30, Mixed Models Analysis

2. Primary Outcome: Changes in Positive Schizophrenia Symptoms
Description: as for outcome 1
Time Frame: Pre-treatment to follow-up, approximately 6 months post end-of-treatment
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive-behavioral Therapy for Psychosis (CBTp) | Supportive Therapy (ST)
Number analyzed (Participants) | 37 | 36
units on a scale
  Baseline | 3.21 (.14) | 3.30 (.14)
  6 Months Post End-of-Tx Follow-up | 3.12 (.15) | 2.78 (.15)
Statistical Analysis 1: Comparison: Cognitive-behavioral Therapy for Psychosis (CBTp) vs Supportive Therapy (ST); Test type: Superiority or Other; p = .09, Mixed Models Analysis

3. Primary Outcome: Changes in Global Social Functioning
Description: Interview rating of overall adaptive functioning rated on a 1-7 scale on the Social Adjust Scale II (Schooler, Hogarty, Weissman:, 1979) with low scores indicating better functioning
  Schooler N, Hogarty G,& Weissman M, (1979). Social Adjustment Scale (SAS) II, in Resource Materials for Community Mental Health Program Evaluators. Edited by Hargreaves W, Attkisson C, Sorenson J. Rockville MD, US Department of Health, Education, and Welfare, 1979, pp 290-303)
Time Frame: Pre-treatment to end of treatment, approximately 6 months post-randomization
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive-behavioral Therapy for Psychosis (CBTp) | Supportive Therapy (ST)
Number analyzed (Participants) | 37 | 37
units on a scale
  Baseline | 5.00 (.12) | 4.80 (.12)
  End of-Active Treatment | 4.78 (.13) | 4.75 (.13)
Statistical Analysis 1: Comparison: Cognitive-behavioral Therapy for Psychosis (CBTp) vs Supportive Therapy (ST); Test type: Superiority or Other; p = .46, Mixed Models Analysis

4. Primary Outcome: Changes in Global Social Functioning
Description: Interview rating of overall adaptive functioning rated on a 1-7 scale on the Social Adjust Scale II (Schooler N, Hogarty G, Weissman M:, 1979) with low scores indicating better functioning
  Schooler N, Hogarty G,& Weissman M, (1979). Social Adjustment Scale (SAS) II, in Resource Materials for Community Mental Health Program Evaluators. Edited by Hargreaves W, Attkisson C, Sorenson J. Rockville MD, US Department of Health, Education, and Welfare, 1979, pp 290-303)
Time Frame: Pre-treatment to follow-up, approximately 6 months post end-of-treatment
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive-behavioral Therapy for Psychosis (CBTp) | Supportive Therapy (ST)
Number analyzed (Participants) | 37 | 36
units on a scale
  Pre-treatment | 5.00 (.12) | 4.80 (.12)
  6 Months Post End-of-Tx Follow-up | 4.63 (.13) | 4.56 (.14)
Statistical Analysis 1: Comparison: Cognitive-behavioral Therapy for Psychosis (CBTp) vs Supportive Therapy (ST); Test type: Superiority or Other; p = .55, Mixed Models Analysis

5. Secondary Outcome: Changes in Distress From Schizophrenia Symptoms
Description: Interview rating of overall preoccupation and distress from hallucinations and delusions rated on the psychotic symptom rating scales (PSYRATS; Haddock, McCarron, Tarrier, & Faragher,; 1999) total score, with a range of 0-85 and low scores indicating less preoccupation and distress
  Haddock, G., McCarron, J., Tarrier, N., & Faragher, E. B. (1999). Scales to measure dimensions of hallucinations and delusions: the psychotic symptom rating scales (PSYRATS). Psychological medicine, 29(04), 879-889.
Time Frame: Pre-treatment to end-of-treatment, approximately 6 months post-randomization
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive-behavioral Therapy for Psychosis (CBTp) | Supportive Therapy (ST)
Number analyzed (Participants) | 37 | 37
units on a scale
  Baseline | 40.79 (2.01) | 40.70 (2.03)
  End of-Active Treatment | 34.45 (2.12) | 36.33 (2.12)
Statistical Analysis 1: Comparison: Cognitive-behavioral Therapy for Psychosis (CBTp) vs Supportive Therapy (ST); Test type: Superiority or Other; p = .50, Mixed Models Analysis

6. Secondary Outcome: Changes in Distress From Schizophrenia Symptoms
Description: as for outcome 5
Time Frame: Pre-treatment to follow-up, approximately 6 months post end-of-treatment
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive-behavioral Therapy for Psychosis (CBTp) | Supportive Therapy (ST)
Number analyzed (Participants) | 37 | 36
units on a scale
  Baseline | 40.79 (2.01) | 40.70 (2.03)
  6 Months Post End of Tx Follow-up | 35.43 (2.15) | 31.48 (2.16)
Statistical Analysis 1: Comparison: Cognitive-behavioral Therapy for Psychosis (CBTp) vs Supportive Therapy (ST); Test type: Superiority or Other; p = .25, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Pre-treatment to 6 month post-treatment follow-up (total 12 months post randomization)
Arm/Group | Cognitive-behavioral Therapy for Psychosis (CBTp) | Supportive Therapy (ST)
Serious Adverse Events (participants affected / at risk) | 11/44 | 12/44
Other Adverse Events (participants affected / at risk) | 0/44 | 0/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive-behavioral Therapy for Psychosis (CBTp) (N=44) | Supportive Therapy (ST) (N=44)
Hospitalization Due to Psychiatric Symptom Exacerbation (Psychiatric disorders) | 6 (6) | 6 (10)
Hospitalization for Cardiac Problems (Cardiac disorders) | 0 (0) | 3 (6)
Hospitalization for Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hospitalization for Fainting (Cardiac disorders) | 1 (1) | 0 (0)
Hospitalization for Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Surgeries (Surgical and medical procedures) | 2 (3) | 1 (1)
Hospitalization for Medication Adjustment (Psychiatric disorders) | 1 (1) | 0 (0)
Hospitalization for Foot Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hospitalization for Dehydration (Endocrine disorders) | 0 (0) | 1 (1)
Hospitalization for Allergic Reaction (General disorders) | 0 (0) | 1 (1)
Hospitalization for Eye Injury (Eye disorders) | 0 (0) | 1 (1)
Hospitalization For Substance Use (Psychiatric disorders) | 1 (2) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes